CLINICAL TRIAL: NCT02107339
Title: Methadone and Hydromorphone For Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director, Clinical Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH14-113
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Hydromorphone Use; Acute Postoperative Pain; Patient Satisfaction; Chronic Persistent Surgical Pain
Keywords: methadone; hydromorphone; acute postoperative pain; chronic persistent surgical pain
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction | interventions — Methadone; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- methadone group (Experimental): Patient will receive methadone 0.2 mg/kg at induction of anesthesia (single dose)
  Interventions: Drug: Methadone
- Hydromorphone group (Active Comparator): Patients will receive hydromorphone 2 mg at the end of the surgical procedure
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Methadone — Methadone 0.2 mg/kg administered at induction of anesthesia
  Arms: methadone group
Drug: Hydromorphone — Hydromorphone 2 mg administered at the conclusion of anesthesia
  Arms: Hydromorphone group

SUMMARY:
Patients undergoing major spinal surgery continue to experience moderate-to-severe pain during the first 2-3 days following the operative procedure. Pain complicates the recovery process, despite the routine practice of using potent opioid analgesics. The primary reason that pain is poorly controlled in patients undergoing major surgery is that most commonly-used opioids only produce analgesia for 2-4 hours. The intermittent use of these drugs results in periods of time when a patient will experience discomfort (at which time a nurse administers more drug or the button on a patient-controlled analgesic (PCA) system is pressed to deliver more medication). The use of a long-acting opioid may be advantageous in the perioperative setting. Methadone is an opioid that has a median duration of analgesia of 24-36 hours. Therefore, a single dose administered in the operating room may reduce the need for pain medication and improve pain control for the first few postoperative days. The aim of this randomized clinical trial is to examine the effect of methadone (compared to hydromorphone) on postoperative pain management in patients undergoing major spine surgery

DETAILED DESCRIPTION:
Patients: 100 patients (ages 18-80) will be enrolled in this clinical trial. All patients presenting for elective posterior lumbar or thoracic spinal fusion surgery will be eligible for enrollment. Patients will be randomized to receive either methadone or hydromorphone on the basis of a computer generated random number table. Patients in each group will receive standard clinical intraoperative doses of either methadone (0.2 mg/kg) or hydromorphone (2 mg). An analysis of patients undergoing posterior lumbar fusion surgery at Evanston Hospital revealed that patients received, on average, approximately 2 mg of hydromorphone intraoperatively. The most commonly used doses of methadone administered in clinical studies have been either 0.2 mg/kg or a dose of 20 mg. Furthermore, these doses also represent dosages which appear to be approximately equipotent. Study medications will be prepared by the pharmacy, and all clinicians will be blinded to group assignment. Two syringes will be prepared for each patient, one which contains the study drug (either methadone 0.2 mg/kg or hydromorphone 2 mg), and the other containing the placebo (saline). If the patient is randomized to the methadone group, a 3 cc syringe containing 0.2 mg/kg of methadone and saline (total volume 3 cc) will be prepared, as well as a 10 cc syringe containing 10 cc of saline (placebo). If the patient is randomized to the hydromorphone group, a 3 cc syringe containing 3 cc of saline (placebo) will be prepared, as well as a 10 cc syringe containing 2 mg of hydromorphone with 9 cc of saline (total volume 10 cc). At induction of anesthesia, the 3 cc syringe containing either 0.2 mg/kg of methadone or placebo will be given over 5 seconds. At the conclusion of surgery, the 10 cc syringe of either hydromorphone or placebo will be titrated slowly per clinician's preference. The administration of all other anesthetic agents will be standardized and reflect the usual practices of anesthesiologists at Evanston Hospital (spine protocol).

Anesthesia will be standardized and include propofol for induction, a propofol and remifentanil infusion for maintenance (plus sevoflurane), and IV acetaminophen 1000 mg during the last 60 minutes of the case.

On arrival to the postanesthesia care unit (PACU), patients will be assessed for pain by PACU nurses per standard protocols. Patients will be evaluated for pain on PACU arrival and then every 15 minutes. Patients will be administered hydromorphone 0.25-0.5 mg for pain, and doses will be repeated until the patient is comfortable (pain < 3 on a scale of 0-10; 0=no pain and 10=worst pain imaginable). The patient will then be connected to a PCA device to deliver pain medication during the remainder of the postoperative period.

All postoperative management will be per standard surgical protocols

Sample Size: The primary end-point of the investigation is amount of hydromorphone used. In a clinical trial by Urban et al. of patients undergoing complex spine surgery using a standard anesthetic, average hydromorphone consumption in the first 24 hours was 27 mg (18). The investigators expect to see at least a 33% reduction in hydromorphone consumption in the methadone group. Group sample sizes of 39 and 39 achieve 91% power to detect a difference of 9.0 between the null hypothesis that both group means are 27.0 and the alternative hypothesis that the mean of group 2 is 18.0 with estimated group standard deviations of 10.0 and 10.0 and with a significance level (alpha) of 0.01000 using a two-sided two-sample t-test. The investigators plan to enroll a total of 100 patients to ensure complete collection of data.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for elective posterior lumbar or thoracic spinal fusion surgery will be eligible for enrollment.

Exclusion Criteria:

1. Preoperative renal failure (defined as a serum creatinine > 2.0 mg/dL.)
2. American Society of Anesthesiologists Physical Status IV or V
3. Pulmonary disease necessitating home oxygen therapy
4. Allergy to methadone or hydromorphone
5. Preoperative recent history of opioid or alcohol abuse
6. Inability to use a PCA device or speak the English language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methadone Group | Hydromorphone Group
Started | 63 | 57
Completed | 62 | 53
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone Group | Hydromorphone Group | Total
Number analyzed (Participants) | 62 | 53 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 34 | 74
  >=65 years | 22 | 19 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.5 [57 to 71] | 60 [45 to 66] | 62 [48 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 32 | 21 | 53
Region of Enrollment [Number; unit: participants]
  United States | 62 | 53 | 115

OUTCOME MEASURES:

1. Primary Outcome: Hydromorphone Use at 24 Hours
Time Frame: Use of hydromorphone at 24 hours
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
milligrams | 4.56 [2.3 to 7.1] | 9.9 [6.45 to 13.2]

2. Secondary Outcome: Hydromorphone Use Second 24 Hours
Time Frame: 24-48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
milligrams | 0.6 [0 to 2.8] | 3.15 [0.75 to 8.2]

3. Secondary Outcome: Hydromorphone Use Third 24 Hours
Time Frame: 48-72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
milligrams | 0 [0 to 0.05] | 0.35 [0 to 3.4]

4. Secondary Outcome: Pain Scores Postanesthesia Care Unit (PACU) Arrival
Description: 11-point verbal rating scale (0=no pain, 10=worst pain imaginable)
Time Frame: First 5 minutes after PACU arrival
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 5 [1 to 7] | 8 [6 to 10]

5. Secondary Outcome: Pain Scores 1 Hour After PACU Arrival
Description: 11-point verbal rating scale (0=no pain, 10=worst pain imaginable)
Time Frame: Pain scores at 60 minutes after PACU admission
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 4 [3 to 6] | 6 [5 to 9]

6. Secondary Outcome: Pain Scores 2 Hours After PACU Arrival
Description: 11-point verbal rating scale (0=no pain, 10=worst pain imaginable)
Time Frame: Pain scores at 120 minutes after PACU admission
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 4 [2 to 4] | 6 [4 to 7]

7. Secondary Outcome: Pain Scores on Postoperative Day One
Description: 11-point verbal rating scale (0=no pain, 10=worst pain imaginable)
Time Frame: Pain scores one day after PACU admission
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 4 [2 to 5] | 5 [3 to 8]

8. Secondary Outcome: Pain Scores on Postoperative Day 2
Description: 11-point verbal rating scale (0=no pain, 10=worst pain imaginable)
Time Frame: Pain scores 48 hours after PACU admission
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 4.56 [2 to 5] | 6 [3.5 to 8]

9. Secondary Outcome: Pain Scores Postoperative Day 3
Description: 11-point verbal rating scale (0=no pain, 10=worst pain imaginable)
Time Frame: Pain scores 72 hours after PACU admission
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 4 [2 to 5] | 5 [3 to 7]

10. Secondary Outcome: Patient Satisfaction Scores
Description: Patient satisfaction with overall pain management will be determined using a 101-point verbal rating scale (0=highly dissatisfied (worst), 100=highly satisfied (best))
Time Frame: Postopertive day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 92.5 [85 to 100] | 80 [70 to 90]

11. Secondary Outcome: Patient Satisfaction Scores
Description: as for outcome 10
Time Frame: postoperative day 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 90 [85 to 100] | 82.5 [70 to 90]

12. Secondary Outcome: Patient Satisfaction Scores
Description: as for outcome 10
Time Frame: Postoperative day 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 62 | 53
units on a scale | 95 [90 to 100] | 90 [77.5 to 95]

13. Secondary Outcome: Chronic Persistent Surgical Pain-Weekly Frequency of Pain
Description: 0=< once per week; 1=once per week; 2=twice per week; 3=daily; 4=constant
Time Frame: One month after surgery
Population: A home postal survey was sent to participants in the clinical trial 1 month after surgery. 41 patients in the methadone group and 34 patients in the hydromorphone group returned the surveys
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 41 | 34
score on a scale | 2 [1 to 3] | 3 [0 to 3]

14. Secondary Outcome: Chronic Persistent Surgical Pain-weekly Frequency of Pain
Description: 0=< once per week; 1=once per week; 2=twice per week; 3=daily; 4=constant
Time Frame: 3 months after surgery
Population: A home postal survey was sent to participants in the clinical trial 3 months after surgery. 38 patients in the methadone group and 27 patients in the hydromorphone group returned the surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 38 | 27
score on a scale | 0 [0 to 3] | 3 [1 to 3]

15. Secondary Outcome: Chronic Persistent Surgical Pain-Weekly Frequency of Pain
Description: 0=< once per week; 1=once per week; 2=twice per week; 3=daily; 4=constant
Time Frame: 6 months after surgery
Population: A home postal survey was sent to participants in the clinical trial 6 months after surgery. 24 patients in the methadone group and 32 patients in the hydromorphone group returned the surveys
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 24 | 32
score on a scale | 0 [0 to 3] | 2 [0 to 3]

16. Secondary Outcome: Chronic Persistent Surgical Pain-Weekly Frequency of Pain
Description: 0=< once per week; 1=once per week; 2=twice per week; 3=daily; 4=constant
Time Frame: 12 months after surgery
Population: A home postal survey was sent to participants in the clinical trial 12 months after surgery. 39 patients in the methadone group and 40 patients in the hydromorphone group returned the surveys
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone Group | Hydromorphone Group
Number analyzed (Participants) | 39 | 40
score on a scale | 0 [0 to 2] | 2 [0 to 3]

ADVERSE EVENTS:
Time Frame: two weeks
Arm/Group | Methadone Group | Hydromorphone Group
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/53
Other Adverse Events (participants affected / at risk) | 0/62 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No